CLINICAL TRIAL: NCT06263712
Title: Differences Between Suicide Attempters and Suicide Ideators. Influence of the Brief Therapy ASSIP on Neuropsychological Correlates and Psychological Process Factors (NePsyASSIP HT) - Project 2
Brief Title: Differences Between Suicide Attempters and Suicide Ideators. Influence of the Brief Therapy Attempted Suicide Short Intervention Program (ASSIP) on Neuropsychological Correlates and Psychological Process Factors - Project 2
Acronym: NePsyAssip HT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-02504 (Project 2)
Record Dates: First submitted 2024-02-08; First posted 2024-02-16 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Inhibitory Control; Self Efficacy; Suicide Ideation; Suicide, Attempted; Locus of Control; Process Factors; Movement Synchrony
MeSH Terms: conditions — Suicide, Attempted | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ASSIP Group (Experimental): Patients in the ASSIP Group will receive 3-4 sessions of the Attempted Suicide Short Intervention Program (ASSIP) which is a specific therapy for patients with a suicide attempt in their personal history. Each ASSIP session takes approximately 50 minutes.
  Interventions: Behavioral: Attempted Suicide Short Intervention Program (ASSIP)
- STAR Group (Active Comparator): Patients in the STAR group will receive the standard of care plus resource interview (STAR) which will be a risk assessment interview, and a non-specific resource focused intervention over three face-to-face sessions. In this resource focused intervention, the sessions are focused on activation of existing resources and the patients' social environment is discussed.
  Interventions: Behavioral: Standard of care plus resource interview group (STAR)

INTERVENTIONS:
Behavioral: Attempted Suicide Short Intervention Program (ASSIP) — The Attempted Suicide Short Intervention Program (ASSIP) is a specific therapy for patients with a suicide attempt in their biography. The brief therapy ASSIP consists of three to four sessions of approximately 50 minutes each.
  Session 1: A narrative interview is conducted, in which the patient is asked to tell her*his personal story which led to the suicidal crisis. The narrative is video-recorded.
  Session 2: Using video-playback of the recorded narrative, patient and therapist explore further details of the suicidal process.
  Session 3: A case conceptualization focusing on the patient's vulnerability and the trigger of the suicidal crisis is formulated in writing. A list of safety strategies for the prevention of future suicidal behavior is developed jointly with the patient.
  Regular letters are sent to patients over a period of 2 years.
  Arms: ASSIP Group
Behavioral: Standard of care plus resource interview group (STAR) — The standard of care plus resource interview group (STAR) will be offered a clinical interview, a risk assessment, and a non-specific resource focused intervention over three face-to-face sessions. In this resource focused intervention, the patient is asked to name her*his resources, describe them, and give examples.
  Arms: STAR Group

SUMMARY:
The present study consists of 3 projects in total and aims to investigate the (neuro-) psychological patterns from suicidal ideation to suicidal behavior as well as the effects and feasibility of ASSIP Home Treatment.

The overall aim of project 2 is to investigate how the (neuro-) psychological patterns are modulated by the Attempted Suicide Short Intervention Program (ASSIP). Therefore, suicide attempters participating in this project 2 will be randomly assigned to either the intervention group ASSIP or a standard care plus resource interview (STAR) group. The ASSIP and STAR interventions take place at the University Hospital of Psychiatry and Psychotherapy Bern (Switzerland).

At the end of the assessment in project 1 participants who reported a history of past suicide attempt (SUAT) will be informed about project 2.

Only if participants agreed to take part in project 2 and have signed the informed consent, they are randomized into two conditions: The ASSIP intervention (ASSIP) versus standard of care plus resource interview (STAR). Participants of both groups will be assessed again 4 weeks and 12 months after their first baseline assessment of project 1.

DETAILED DESCRIPTION:
Purpose and aims:

The present study consists of 3 projects in total and aims to investigate the (neuro-) psychological patterns from suicidal ideation to suicidal behavior as well as the effects and feasibility of ASSIP Home Treatment.

After the cross-sectional study in project 1 determining the (neuro-) psychological patterns between suicide ideators (SUID) and suicide attempters, in project 2, the aim is to learn more about the (neuro-) psychological patterns and how they are modulated by a suicide-specific brief intervention ASSIP that was proven to be effective. In addition to the (neuro-) psychological assessment, longitudinal process factors are examined by comparing an ASSIP intervention group to a group of standard care plus resource interview (STAR). The STAR intervention refers to the usual and customary practices within the field, including suicide risk assessment, a non-specific resource focused intervention and if necessary, further outpatient or inpatient treatment.

Background:

In Switzerland, approximately three people die by suicide every day and suicide attempts exceed this number by far. As a previous suicide attempt is one of the strongest predictors for a completed suicide, it is of utmost importance to identify the people at risk. However, research has shown that traditional risk factors (e.g., depression, psychiatric disorder, etc.) reliably predict suicide ideation but poorly predict suicidal behavior. Furthermore, while effective suicide-specific interventions exist, up to 50% of the suicide attempters reject the recommended treatment and around 60% discontinue treatment after one session. Hence, a different approach is required. In this study, three projects will be conducted. Project 1 aims is to identify the (neuro-) psychological patterns of suicidal attempters by comparing between the following four different groups:

1) patients with a prior suicide attempt (SUAT) 2) patients with no prior suicide attempt, but suicidal ideation (SUID) 3) a general patient group (CLIN), and 4) a healthy control group (HLTH).

Project 2 aims to investigate how these patterns are modulated by the efficacious brief therapy ASSIP. In project 3, the feasibility, effects and cost-effectiveness of the ASSIP Home Treatment will be investigated.

Study design of project 2:

A longitudinal analysis over 12 months will only be conducted for the SUAT group. SUAT who participated in project 1 will be asked whether they also wish to participate in project 2. If they agree, they will be randomly assigned to either the intervention group ASSIP or STAR group to understand the influence of the brief ASSIP on (neuro-) psychological correlates in suicide attempters. The brief therapy ASSIP and STAR will take place at the University Hospital of Psychiatry and Psychotherapy Bern (Switzerland). Participants in project 2 will be assessed at 4 weeks, and 12 months after the first assessment which was conducted within project 1 and participants will be assessed on several process factors after each ASSIP or STAR session.

ELIGIBILITY:
Inclusion Criteria for Project 2:

Subjects fulfilling the following inclusion criteria are eligible for the study:

* Informed consent as documented by signature
* Age ≥ 18 years
* At least one previous suicide attempt
* Willingness to attend the ASSIP brief therapy
* Owns a smartphone

Exclusion Criteria for Project 2:

The presence of any one of the following exclusion criteria will lead to exclusion of the subject:

* Serious cognitive impairment
* Any psychotic disorder
* Any current medication, which substantially impairs the attention span, reaction, rate or any other relevant cognitive functions
* Inability to follow the procedures of the study (e.g., insufficient mastery of the German language, previous enrolment into the current study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Differences in Inhibitory Control | The assessment takes place 1 day to 1 week after informed consent (t0).
  The Go/No-Go task is a cognitive task to assess an individual's ability to inhibit a prepotent response. It is used to measure impulse control and response inhibition. The task requires participants to respond ("Go" response) to one type of stimulus and to withhold or inhibit their response ("No-Go" response) to another type of stimulus. The Go/No-Go task yields measures such as reaction time, accuracy, and the ability to inhibit responses. Reaction times can vary widely, and accuracy is often expressed as a percentage of correct responses. Lower reaction times and higher accuracy in withholding responses (No-Go trials) indicate better inhibitory control and cognitive performance.
Differences in Inhibitory Control | The assessment takes place after the completion of the 3/4 ASSIP or STAR therapy sessions (t1), i.e. approximately 4 weeks after the baseline assessment.
  The Go/No-Go task is a cognitive task to assess an individual's ability to inhibit a prepotent response. It is used to measure impulse control and response inhibition. The task requires participants to respond ("Go" response) to one type of stimulus and to withhold or inhibit their response ("No-Go" response) to another type of stimulus. The Go/No-Go task yields measures such as reaction time, accuracy, and the ability to inhibit responses. Reaction times can vary widely, and accuracy is often expressed as a percentage of correct responses. Lower reaction times and higher accuracy in withholding responses (No-Go trials) indicate better inhibitory control and cognitive performance.
Differences in Inhibitory Control | The assessment takes place 12 months after the baseline assessment (t2).
  The Go/No-Go task is a cognitive task to assess an individual's ability to inhibit a prepotent response. It is used to measure impulse control and response inhibition. The task requires participants to respond ("Go" response) to one type of stimulus and to withhold or inhibit their response ("No-Go" response) to another type of stimulus. The Go/No-Go task yields measures such as reaction time, accuracy, and the ability to inhibit responses. Reaction times can vary widely, and accuracy is often expressed as a percentage of correct responses. Lower reaction times and higher accuracy in withholding responses (No-Go trials) indicate better inhibitory control and cognitive performance.

SECONDARY OUTCOMES:
Movement analyses | The assessment takes place at all 3 sessions of ASSIP or STAR, up to 1 month.
  To assess nonverbal synchrony between patient and therapist, all ASSIP and STAR sessions are recorded by video cameras. The video recordings of the ASSIP sessions are subjected to Motion Energy Analysis (MEA), an objective, automatized assessment of participant's movement dynamics. MEA uses an image-differencing algorithm common to the context of computer vision, and well suited for the quantification of movement dynamics from two-dimensional recordings.The MEA program provides four continuous time-series representing the amount of movement in the head and gesture regions of both the patient and the ASSIP therapist. Based on these time-series of objective movement-quantification, a measure of nonverbal synchrony is carried out by a specific cross-correlation function.
Selective Attention and Interference Control | The assessment takes place 1 day to 1 week after informed consent (t0); after the completion of the 3/4 ASSIP or STAR sessions, i.e. approximately 4 weeks after the baseline assessment (t1); 12 months after the baseline assessment (t2).
  The Stroop task is a cognitive psychology test that evaluates an individual's ability to selectively attend to information while inhibiting interference from irrelevant stimuli. The Stroop task measures the time taken to complete tasks and the accuracy of responses. The primary measures are the time taken to complete the task and the number of errors. Lower completion times and fewer errors indicate better cognitive control and attentional focus. Lower scores (faster completion times and fewer errors) are associated with better outcomes, reflecting more efficient cognitive processing and interference control. Higher scores, if used to quantify errors or time taken, are associated with a worse outcome, indicating greater interference and potentially reduced cognitive control.
General Sense of Self-Efficacy | The assessment takes place 1 day to 1 week after informed consent (t0); after the completion of the 3/4 ASSIP or STAR sessions, i.e. approximately 4 weeks after the baseline assessment (t1); 12 months after the baseline assessment (t2).
  The General Self-Efficacy Scale (GSE) is a 10-item self-report questionnaire to assess the general sense of self-efficacy. Items are rated from 1 (do not agree) to 4 (totally agree). A higher score indicates a stronger belief in one's ability to cope with and navigate different situations.
Locus of control | The assessment takes place 1 day to 1 week after informed consent (t0); after the completion of the 3/4 ASSIP or STAR sessions, i.e. approximately 4 weeks after the baseline assessment (t1); 12 months after the baseline assessment (t2).
  The Internal-External Locus of Control Short Scale-4 (IE-4) is a brief measure designed to assess an individual's locus of control orientation. Locus of control refers to the extent to which individuals believe they control events in their lives. The IE-4 is typically scored by summing the responses to its four items, each rated on a Likert scale. The possible score range is determined by the specific scoring method researchers or practitioners use. The scores may range from 4 to 16, depending on the scoring system employed. Higher scores on the IE-4 may suggest a more internal locus of control, indicating a belief that one has control over their life events. Lower scores may indicate a more external locus of control, suggesting a belief that external factors or luck play a significant role in life events.
Psychological Pain | The assessment takes place 1 day to 1 week after informed consent (t0); after the completion of the 3/4 ASSIP or STAR sessions, i.e. approximately 4 weeks after the baseline assessment (t1); 12 months after the baseline assessment (t2).
  The Mee-Bunney Psychological Pain Assessment Scale (MBPPAS) is a 10-item self-report scale to assess intensity and frequency of psychological pain. Psychological pain is defined as an experience of unbearable agony which can be linked to a psychiatric disorder.
Suicidal ideation and behavior | The assessment takes place 1 day to 1 week after informed consent (t0); after the completion of the 3/4 ASSIP or STAR sessions, i.e. approximately 4 weeks after the baseline assessment (t1); 12 months after the baseline assessment (t2).
  The Self-Injurious Thoughts and Behaviors Interview (SITBI) is a structured interview that assesses the presence, frequency, and characteristics of a wide range of self-injurious thoughts and behaviors, including suicidal ideation, suicide plans, suicide gestures, suicide attempts, and nonsuicidal self-injury. We will draw on selected questions from this interview and apply them in the form of a questionnaire.
Suicidal ideation | The assessment takes place 1 day to 1 week after informed consent (t0); after the completion of the 3/4 ASSIP or STAR sessions, i.e. approximately 4 weeks after the baseline assessment (t1); 12 months after the baseline assessment (t2).
  The Beck Scale for Suicide Ideation (BSS) is a self-report questionnaire with 21 items. The BSS measures the ideation (suicidal thoughts, plans and suicidal feeling) of suicide.

OTHER OUTCOMES:
Mental abilities like attention, working memory and visuomotor speed as well as mental flexibility | The assessment takes place 1 day to 1 week after informed consent (t0); after the completion of the 3/4 ASSIP or STAR sessions, i.e. approximately 4 weeks after the baseline assessment (t1); 12 months after the baseline assessment (t2).
  The Trail Making Test (TMT-A/B) is a neuropsychological test that assesses visual attention and task-switching abilities. It consists of two parts (Part A and Part B) and measures the time taken to complete each part. The score is typically represented as the time (in seconds) taken to complete the task. Lower scores (faster completion times) are generally considered better outcomes, indicating more efficient visual attention, processing speed, and cognitive flexibility. Higher scores (longer completion times) may suggest difficulties in these cognitive domains and are typically associated with worse outcomes.
Sociodemographic data | The assessment takes place 1 day to 1 week after informed consent (t0); after the completion of the 3/4 ASSIP or STAR sessions, i.e. approximately 4 weeks after the baseline assessment (t1); 12 months after the baseline assessment (t2).
  The Sociodemographic Questionnaire (DEMO) is a 30-item questionnaire that was developed to collect sociodemographic (e.g., gender, socioeconomic status, professional status, relationship satisfaction) and health-related data (e.g., medication, inpatient and outpatient treatment).
Diagnostic and Statistical Manual 5 (DSM-V) and International Classification of Diseases 10 (ICD-10) psychiatric disorders | The assessment takes place 1 day to 1 week after informed consent (t0).
  The Mini-DIPS is a short, structured clinical interview for diagnosing mental disorders and is based on the DIPS-OA. The Mini-DIPS allows for a quick yet reliable diagnosis. It is applicable in adulthood and captures lifetime diagnoses, current and past diagnoses, based on the criteria of DSM-5 and ICD-10. The Mini-DIPS covers the mental disorders most commonly observed in clinical settings.
Depressive symptoms | The assessment takes place 1 day to 1 week after informed consent (t0); after the completion of the 3/4 ASSIP or STAR sessions, i.e. approximately 4 weeks after the baseline assessment (t1); 12 months after the baseline assessment (t2).
  The Beck Depression Inventory (BDI-II) is a self-assessment questionnaire and contains 21 items which assess the severity of depressive symptoms. A participant's score is calculated by summing up the scores from each item. The total score ranges from 0 to 63. Values between 0 and 11 lie within the norm, between 11 and 17 moderate depressive symptoms and a total score up to 18 is assessed as a clinically relevant depressive disorder.
Loneliness | The assessment takes place 1 day to 1 week after informed consent (t0); after the completion of the 3/4 ASSIP or STAR sessions, i.e. approximately 4 weeks after the baseline assessment (t1); 12 months after the baseline assessment (t2).
  The Three-Item UCLA (University of California, Los Angeles) Loneliness Scale is a short questionnaire with three items from the Revised UCLA Loneliness Scale (R-UCLA). These items can be rated from 1 (hardly ever) to 3 (often). A higher score indicates a higher level of perceived loneliness. The scale is designed to measure subjective feelings of loneliness, so individuals who score higher on the UCLA Loneliness Scale report more frequent experiences of loneliness and social isolation.
Therapeutic Alliance | The assessment takes place at all 3 sessions of ASSIP or STAR, up to 1 month.
  The Working Alliance Inventory - short revised (WAI-SR) in German is an empirically validated and economic instrument to assess the therapeutic alliance.
Therapeutic change | The assessment takes place after the third session of ASSIP or STAR (week 3).
  The Bochum Change Questionnaire 2000 (BVB-2000) is a direct self-report assessment for therapeutic change.
Therapeutic outcomes | The assessment takes place at all 3 sessions of ASSIP or STAR, up to 1 month.
  The Questionnaire for the evaluation of psychotherapy processes (FEP-2) assesses four dimensions of therapeutic outcomes (Well-Being, General symptoms, Incongruence and Interpersonal problems).
Adherence and Competence | The assessment takes place at all 3 sessions of ASSIP or STAR, up to 1 month.
  Adherence and Competence Scales, element 1-5 (ACS). The ACS scales were developed using the ASSIP criteria.
Physiologically Experienced Emotional Distress and Arousal | The assessment takes place 1 day to 1 week after informed consent (t0); after the completion of the 3/4 ASSIP or STAR sessions, i.e. approximately 4 weeks after the baseline assessment (t1); 12 months after the baseline assessment (t2).
  Electrodermal activity (EDA), also known as skin conductance or galvanic skin response, is a valuable physiological marker in suicide research. EDA measures the skin's electrical conductance, reflecting sympathetic nervous system activity. Suicidal individuals often experience heightened emotional distress and arousal, challenging assessment via self-reports alone. EDA offers an objective, non-invasive means to quantify this emotional response, with distinct patterns observed in those at risk of suicide.
Ecological Momentary Assesment | Always three days before and three days after each ASSIP/STAR therapy session. Starts approximately 1 week after the informed consent and finishes approximately 4 weeks after the informed consent.
  Real-time measurement of patients' risk factors using a phone app M-path. A 14-items questionnaire which is filled out 5 times a day.
Attention and Concentration Abilities | The assessment takes place 1 day to 1 week after informed consent (t0); after the completion of the 3/4 ASSIP or STAR sessions, i.e. approximately 4 weeks after the baseline assessment (t1); 12 months after the baseline assessment (t2).
  The D2 Test of Attention and Concentration is a neuropsychological test used to assess selective and sustained attention. It is employed to evaluate an individual's visual scanning, concentration, and information processing speed. The D2 Test involves scoring based on the number of correctly marked items minus the number of errors. The scoring method considers both the quantity and accuracy of responses. The goal is to mark as many target items as possible within a specified time limit while avoiding errors. A higher score is considered a better outcome, indicating more correct responses and effective attention and concentration.
Dissociative Experience | The assessment takes place 1 day to 1 week after informed consent (t0); after the completion of the 3/4 ASSIP or STAR sessions, i.e. approximately 4 weeks after the baseline assessment (t1); 12 months after the baseline assessment (t2).
  The German Dissociation-Tension Scale - 4 (DSS-4) is a four-item brief self-report instrument to assess dissociation. It was developed based on the DSS-acute, a longer scale to measure dissociative symptoms. The four DSS-4 items assess somatic and psychological dissociation and each item is rated on a 10-point Likert scale ranging from "not present" = 0 to "very strong" = 9. Based on the DSS-4, a dissociation score per participant is calculated as the mean of the four items.
Motivational Incongruence | The assessment takes place 1 day to 1 week after informed consent (t0); after the completion of the 3/4 ASSIP or STAR sessions, i.e. approximately 4 weeks after the baseline assessment (t1); 12 months after the baseline assessment (t2).
  The Incongruence Questionnaire (INK) measures unsatisfactory realization of motivational goals, whereas the personal relevance of motivation is measured in the FAMOS. The questionnaire INK assesses the realization of approach and avoidance goals on 14 and 9 scales, respectively, with a total of 94 items. Each item to assess approach goals is assessed on a five-point Likert scale. For each scale, the mean value of the corresponding item values must be determined. In addition, it is possible to calculate three composite scales: 1) incongruence with avoidance goals; 2) incongruence with approach goals; and 3) total incongruence.
Motivational Goals | The assessment takes place 1 day to 1 week after informed consent (t0).
  The Questionnaire for the Analysis of Motivational Schemas (FAMOS) assesses the motivational goals of psychotherapy in terms of central components of motivational schemas in self-report format. The questionnaire FAMOS assesses motivational goals as approach goals on 14 scales and avoidance goals on 9 scales, with a total of 94 items. Each item is rated on a five-point Likert scale. For each scale, the scale mean of the corresponding items is calculated. In addition, three summary values can be calculated: 1) total value for approach goals; 2) total value for avoidance goals; and 3) the ratio of avoidance to approach goals.
Suicide-Related Coping | The assessment takes place 1 day to 1 week after informed consent (t0); after the completion of the 3/4 ASSIP or STAR sessions, i.e. approximately 4 weeks after the baseline assessment (t1); 12 months after the baseline assessment (t2).
  Coping with suicidal ideation and behavior will be assessed with the Suicide-Related Coping Scale (SRCS). The self-report scale SCRS consists of 17 items, with each rated on a five-point Likert scale from "strongly disagree" = 0 to "strongly agree" = 4. A total SRCS sum score is calculated by inverting the negatively worded items and then summing the 17 items. A higher sum score indicates better suicide-related coping.
Alcohol Use Screening | The assessment takes place 1 day to 1 week after informed consent.
  The Alcohol Use Disorders Identification Test (AUDIT-C) is an alcohol screen that is used to identify patients who are hazardous drinkers or who may have an active alcohol use disorder. The minimum score (for non-drinkers) is 0, and the maximum possible score is 12. The higher the AUDIT-C score, the more likely it is that the patient's drinking is affecting their health and safety.

CONTACTS AND LOCATIONS:
Overall Officials: Anja C. Gysin-Maillart, PhD, Principal Investigator — University of Bern, University Hospital of Psychiatry, Translational Research Center
Locations (1):
- University Hospital of Psychiatry and Psychotherapy, University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peter, C. and A. Tuch, Suizidgedanken und Suizidversuche in der Schweizer Bevölkerung. Obsan Bulletin. Vol. 7. 2019, Nêuchatel. 2019.
- [Background] Bostwick JM, Pabbati C, Geske JR, McKean AJ. Suicide Attempt as a Risk Factor for Completed Suicide: Even More Lethal Than We Knew. Am J Psychiatry. 2016 Nov 1;173(11):1094-1100. doi: 10.1176/appi.ajp.2016.15070854. Epub 2016 Aug 13. PMID 27523496
- [Background] Ystgaard M, Arensman E, Hawton K, Madge N, van Heeringen K, Hewitt A, de Wilde EJ, De Leo D, Fekete S. Deliberate self-harm in adolescents: comparison between those who receive help following self-harm and those who do not. J Adolesc. 2009 Aug;32(4):875-91. doi: 10.1016/j.adolescence.2008.10.010. Epub 2008 Nov 22. PMID 19028399
- [Background] Klonsky ED, May A. Rethinking impulsivity in suicide. Suicide Life Threat Behav. 2010 Dec;40(6):612-9. doi: 10.1521/suli.2010.40.6.612. PMID 21198330
- [Background] May, A.M. and E.D. Klonsky, What distinguishes suicide attempters from suicide ideators? A meta-analysis of potential factors. Clinical Psychology: Science and Practice, 2016. 23(1): p. 5.
- [Background] Lizardi D, Stanley B. Treatment engagement: a neglected aspect in the psychiatric care of suicidal patients. Psychiatr Serv. 2010 Dec;61(12):1183-91. doi: 10.1176/ps.2010.61.12.1183. PMID 21123401
- [Background] Schiepek, G., Ressourcenorientierung und Ressourcendiagnostik in der Psychotherapie. 2003.
- [Background] Gysin-Maillart, A., ASSIP - Kurztherapie nach Suizidversuch. Attempted Sucide Short Intervention Program. 2. Aufl. ed. 2021, Bern: Hogrefe.
- [Background] Smith JL, Mattick RP, Jamadar SD, Iredale JM. Deficits in behavioural inhibition in substance abuse and addiction: a meta-analysis. Drug Alcohol Depend. 2014 Dec 1;145:1-33. doi: 10.1016/j.drugalcdep.2014.08.009. Epub 2014 Aug 24. PMID 25195081
- [Background] Nock MK, Hwang I, Sampson NA, Kessler RC. Mental disorders, comorbidity and suicidal behavior: results from the National Comorbidity Survey Replication. Mol Psychiatry. 2010 Aug;15(8):868-76. doi: 10.1038/mp.2009.29. Epub 2009 Mar 31. PMID 19337207
- [Background] Rath D, Hallensleben N, Glaesmer H, Spangenberg L, Strauss M, Kersting A, Teismann T, Forkmann T. [Implicit Associations with Death: First Validation of the German Version of the Suicide Implicit Association Test (Suicide IAT)]. Psychother Psychosom Med Psychol. 2018 Mar;68(3-4):109-117. doi: 10.1055/s-0043-105070. Epub 2017 Jun 29. German. PMID 28718868
- [Background] Ramseyer F, Tschacher W. Nonverbal synchrony in psychotherapy: coordinated body movement reflects relationship quality and outcome. J Consult Clin Psychol. 2011 Jun;79(3):284-95. doi: 10.1037/a0023419. PMID 21639608
- [Background] MacLeod CM, MacDonald PA. Interdimensional interference in the Stroop effect: uncovering the cognitive and neural anatomy of attention. Trends Cogn Sci. 2000 Oct 1;4(10):383-391. doi: 10.1016/s1364-6613(00)01530-8. PMID 11025281
- [Background] Reitan, R.M. and D. Wolfson, Category Test and Trail Making Test as measures of frontal lobe functions. The Clinical Neuropsychologist, 1995. 9(1): p. 50-56.
- [Background] Schwarzer, R. and M. Jerusalem, Skala zur allgemeinen Selbstwirksamkeitserwartung. 1999, Berlin: Freie Universität Berlin. 2013.
- [Background] Kovaleva, A., et al., Eine Kurzskala zur Messung von Kontrollüberzeugung: Die Skala Internale-Externale-Kontrollüberzeugung-4 (IE-4). 2012.
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] Beck AT, Steer RA, Ranieri WF. Scale for Suicide Ideation: psychometric properties of a self-report version. J Clin Psychol. 1988 Jul;44(4):499-505. doi: 10.1002/1097-4679(198807)44:43.0.co;2-6. PMID 3170753
- [Background] Mee S, Bunney BG, Bunney WE, Hetrick W, Potkin SG, Reist C. Assessment of psychological pain in major depressive episodes. J Psychiatr Res. 2011 Nov;45(11):1504-10. doi: 10.1016/j.jpsychires.2011.06.011. Epub 2011 Aug 9. PMID 21831397
- [Background] Hautzinger, M., et al., Beck-depressions-inventar (BDI). Bearbeitung der deutschen Ausgabe. Testhandbuch. Bern: Huber, 1994.
- [Background] Hughes ME, Waite LJ, Hawkley LC, Cacioppo JT. A Short Scale for Measuring Loneliness in Large Surveys: Results From Two Population-Based Studies. Res Aging. 2004;26(6):655-672. doi: 10.1177/0164027504268574. PMID 18504506
- [Background] Munder T, Wilmers F, Leonhart R, Linster HW, Barth J. Working Alliance Inventory-Short Revised (WAI-SR): psychometric properties in outpatients and inpatients. Clin Psychol Psychother. 2010 May-Jun;17(3):231-9. doi: 10.1002/cpp.658. PMID 20013760
- [Background] Willutzki, U., et al., Direkte Veränderungsmessung in der Psychotherapie. Zeitschrift für Klinische Psychologie und Psychotherapie, 2013.
- [Background] Hasler G, Klaghofer R, Buddeberg C. [The University of Rhode Island Change Assessment Scale (URICA)]. Psychother Psychosom Med Psychol. 2003 Sep-Oct;53(9-10):406-11. doi: 10.1055/s-2003-42172. German. PMID 14528410
- [Background] Gysin-Maillart, Michel, Conner, Westrin and Ehnvall (in progress).
- [Background] Russell D, Peplau LA, Cutrona CE. The revised UCLA Loneliness Scale: concurrent and discriminant validity evidence. J Pers Soc Psychol. 1980 Sep;39(3):472-80. doi: 10.1037//0022-3514.39.3.472. PMID 7431205
- [Background] Klonsky, E.D. and A.M. May, The three-step theory (3ST): A new theory of suicide rooted in the
- [Background] Teismann T, et al., Skala Suizidales Erleben und Verhalten (SSEV). Diagnostica. 2021; 67(3): 115-125.
- [Background] Lutz W, Böhnke JR. Der